CLINICAL TRIAL: NCT06547008
Title: Army-Suicide Prevention Research on Implementation in the National Guard (Army-SPRING)
Brief Title: Army-SPRING Army-Suicide Prevention Research
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 855941
Record Dates: First submitted 2024-07-11; First posted 2024-08-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Suicide
Keywords: suicide; military
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Army-SPRING (Experimental): Army-SPRING includes a package of implementation options to support implementation of suicide prevention duties
  Interventions: Behavioral: Army-SPRING
- Risk Reduction Group (Control) (Placebo Comparator): Risk Reduction Group is a mandated training from National Guard Service members
  Interventions: Behavioral: Risk Reduction Group (Control)

INTERVENTIONS:
Behavioral: Army-SPRING — Army-SPRING includes a package of implementation options to support implementation of suicide prevention duties
  Arms: Army-SPRING
Behavioral: Risk Reduction Group (Control) — Risk Reduction Group is a mandated training from National Guard Service members
  Arms: Risk Reduction Group (Control)

SUMMARY:
Every unit in the Connecticut Army National Guard has a Suicide Intervention Officer to provide suicide intervention education awareness for their unit, monitor for soldiers in crisis and connect soldiers with helping resources and agencies. Suicide Intervention Officers need support in this difficult role, yet there is limited guidance on how to help them. This study will shed light on how to support Suicide Intervention Officers and whether this support results in reduced suicide risk in their units.

DETAILED DESCRIPTION:
Attachment 4: Lay Abstract Objective 1: The first objective is to spend 6 months collecting feedback from Army National Guard Soldiers and their family, the religious affairs team, and leadership on how best to reduce risk for suicide. We will also collect feedback from Suicide Intervention Officers, who are appointed to reduce risk for suicide in their unit, about how to support these officers in their important work.

Objective 2: The second objective is to compare two strategies to support Suicide Intervention Officers as they work closely with soldiers to reduce their risk for suicide. The 47 Suicide Intervention Officers in the Connecticut Army National Guard will be randomly assigned (like the flip of a coin) to one of two groups. The first group will attend an extra training (Control Group). The second group will become part of a community focused on reducing suicide risk, including access to online forums to support them in their work, support in leading Battle Drills focused on suicide prevention, and additional training and consultation (Army-SPRING Group). Chaplains/religious affairs specialists will also receive the Army-SPRING group training, but will not be randomized since there are only 5 total Chaplains and 5 religious affairs specialists.

Objective 3: The third objective is to study whether soldiers with Suicide Intervention Officers in the Army-SPRING Group (described in objective 2) report lower rates of suicide ideation and attempts than the Control Group.

Rationale: Every unit in the Connecticut Army National Guard has a Suicide Intervention Officer to provide suicide intervention education awareness for their unit, monitor for soldiers in crisis and connect soldiers with helping resources and agencies. Suicide Intervention Officers need support in this difficult role, yet there is limited guidance on how to help them. This study will shed light on how to support Suicide Intervention Officers and whether this support results in reduced suicide risk in their units.

CBPR Approach and Implementation: We have formed a community advisory board that includes Veterans of Army National Guard units in other states (Pennsylvania); Veterans of the Army with employment as a civilian in the Marines, Chaplains in the Connecticut National Guard on the Air Force (who are intimately familiar with the needs at CT but who are not employees of the Army National Guard), and members of the Suicide Prevention Task force. We have asked for their feedback on the design of the study and will meet with them monthly for the three months and then quarterly thereafter.

FY23 TBIPHRP HSRA Focus Area: This project relates to the Prevent and Assess area of encouragement namely: "Development, evaluation, and implementation of crosscutting prevention approaches targeting upstream factors or leveraging communities and peers to address multiple adverse outcomes such as suicide." Types of Patients Helped by the Research and How it will Help Them: This research will help Army National Guard Soldiers, who are at higher risk for suicide than Active Duty service members. It will help them by supporting Suicide Intervention Officers as they work to reduce risk for suicide among soldiers.

Potential clinical applications, Benefits and Risks: The clinical application is a strategy to support Suicide Intervention Officers, which could benefit soldiers in reducing their suicide risk.

Projected timeline: 4 years, including 6 months of preparatory work with our community advisory board, who will also provide input throughout.

Health and well-being of Service Members: This will help the health and well-being of service members by reducing their risk for suicide. It will help Suicide Intervention Officers by improving their confidence in supporting soldiers who are struggling with suicide risk. It will help Chaplains/Religious affairs specialists who regularly desire more training in suicide prevention and who are a well-used source of support for soldiers at risk.

ELIGIBILITY:
Inclusion Criteria:

* Serving as an SIO or chaplain/religious affairs specialist for a unit of the CTARNG
* Willing to provide informed consent.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Reach - Self | Year 1
  Use of suicide prevention services for self, URI-3 item 75
Reach - Intervening for others | Year 1
  Use of suicide prevention services for buddy, URI-3 item 74
Reach - Interactions with soldiers involving discussions about suicide risk | Weekly for 1 year
  Number of soldier interactions reporting suicide risk/Total number of interactions with soldiers

SECONDARY OUTCOMES:
Suicidal ideation | Year 1
  URI-3 item 15
Suicide plans: | Year 1
  URI-3 item 15a
Suicide attempts | Year 1
  URI-3 item 15b
Adoption | Up to 24 months
  Suicide intervention officer willingness to initiate all SIO duties; This will be operationalized as the total number of SIOs who reported willingness to complete all their suicide prevention-related activities
Implementation | Up to 24 months
  Fidelity to all assigned suicide intervention officer duties; Fidelity will be assessed using self-report by the SIO, including the following questions: 1) Does your battalion know that you are their SIO?; and 2) Have you completed any trainings related to suicide prevention with your battalion? Finally, among SIOs randomized to ARMY-SPRING, we will assess their fidelity of leading the battle drills in a manner consistent with suicide prevention principals.
Acceptability | Up to 24 months
  Acceptability of Intervention Measure (AIM)
Appropriateness | Up to 24 months
  Intervention appropriateness measure (IAM)
Qualitative Interviews | Up to 24 months
  Qualitative Interviews (Acceptability, appropriateness, climate, etc.)

OTHER OUTCOMES:
Intentions, attitudes, norms | Baseline, quarterly, year 1, year 2
  Theory of Planned Behavior Questionnaire
Organizational culture | Baseline, quarterly, year 1, year 2
  We use the support subscale of the Implementation Leadership Scale to assess how leadership influences implementation outcomes. Organizational culture measures the culture and climate in their battalion, feasibility and acceptability of implementing suicide prevention tasks
Maintenance | Up to 24 months
  Suicidal ideation: URI-3 item 15; Suicide plans: URI-3 item 15a

CONTACTS AND LOCATIONS:
Overall Officials: Lily Brown, PhD, Principal Investigator — University of Pennsylvania; Ashley Hagaman, PhD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Connecticut Army National Guard, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Center for the Treatment and Study of Anxiety, University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
We will upload data into the NIMH Data Archives every 6 months.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Each 6 months once official data collection begins.
Access Criteria: Determined by the NIMH
URL: https://nda.nih.gov/